CLINICAL TRIAL: NCT01185184
Title: A Phase 1, Randomized, 3-Period, Open Label, Single Dose, Cross Over Study To Evaluate The Pharmacokinetics And Safety Of Two Controlled Release Formulations Of CP-690,550
Brief Title: Pharmacokinetics And Safety Study Of Two CP-690,550 Controlled Release Formulation Following Single Dose In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A3921113
Record Dates: First submitted 2010-08-18; First posted 2010-08-19 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Healthy
Keywords: Relative bioavailability; controlled release; Phase 1; CP-690; 550
MeSH Terms: interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Subjects will receive in random order, the immediate release tablet containing 10 mg of CP-690,550 and two different controlled-release capsules containing 20 mg of CP-690,550.
  Interventions: Drug: CP-690,550

INTERVENTIONS:
Drug: CP-690,550 — Single doses separated by a minimum of 72 hour washout between treatments

SUMMARY:
This study will explore the drug behavior and safety following single dose of two 20 milligram CP-690,550 osmotic capsules in 12 healthy volunteers. These will be compared to a 10 milligram immediate release tablet, using a 3 way crossover design.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease.
* Clinically significant infections within the past 3 months.

Ages: 21 Months to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2010-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters: AUCinf(dn), Frel and Cmax(dn) of CP-690,550 | 36 hours

SECONDARY OUTCOMES:
Pharmacokinetic parameters: AUCinf, AUClast, AUClast(dn), Cmax, Tmax, t½, C12h, C24h of CP-690,550 | 9 days
Safety: laboratory tests, adverse events reporting, ECG and vital signs | 9 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921113&StudyName=Pharmacokinetics%20And%20Safety%20Study%20Of%20Two%20CP-690%2C550%20Controlled%20Release%20Formulation%20Following%20Single%20Dose%20In%20Healthy%20Volunteers